CLINICAL TRIAL: NCT01460069
Title: The Effect of GLP-1 in Psoriasis
Brief Title: The Effect of Glucagon Like Peptide (GLP)-1 in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Annesofie Faurschou (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Annesofie Faurschou, MD PhD - Resident in dermatology, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-000571-13
Record Dates: First submitted 2011-10-18; First posted 2011-10-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Psoriasis
Keywords: psoriasis; liraglutide; morbidity; PASI; DLQI
MeSH Terms: conditions — Psoriasis | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Victoza treatment (Active Comparator)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator): The placebo pens contain saline and are administered in the same way and volume as Victoza. The placebo pens are specially prepared for this study and will be used in the study only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: liraglutide — Victoza® is supplied in pens for injection containing 18 mg of the GLP-1 agonist liraglutide in 3 mL sterile water with disodiumphosphate and propylenglycol, and phenol for conservation (pH 8.15). Commercial pens will be used and the information given in the packaging will be applicable. The initial daily dose will be 0.6 mg for one week, 1.2 mg the following week and then 1.8 mg for the remaining treatment period. The injection is administered once daily in the morning. The maximal plasma concentration is reached 8-12 hours after subcutaneous injection. The half-life in plasma is approximately 13 hours. The duration of effect is 24 hours.
  Arms: Victoza treatment
Drug: Placebo — The placebo pens contain saline and are administered in the same way and volume as (liraglutide) Victoza. The placebo pens are specially prepared for this study and will be used in the study only.
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the effect of the GLP-1 analogue Victoza® on psoriasis in a double-blinded, randomized placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians above 18 years of age
* Plaque psoriasis
* PASI score >10
* No treatment or stable treatment of psoriasis during at least 3 months before inclusion
* Steady weight through 3 months with a body mass index (BMI) above 27 kg/m2
* Normal blood pressure
* Spiral or hormonal birth control for fertile women during the entire treatment period and at least 3 days after the end of the treatment period (~5 times the plasma half-life)

Exclusion Criteria:

* Psoriasis arthritis
* Fasting plasma glucose > 7.5 mmol/L or HbA1c > 7.5%
* Type 1 diabetes
* Treatment for type 2 diabetes with GLP-1-based medicine (DDP-4-inhibitors or GLP-1-receptor-agonists)
* Heart failure, NYHA class III-IV
* Uraemia, end-stage renal disease, or any other cause of impaired renal function with s-creatinine >150 µM and/or albuminuria
* Liver disease (alanine amino transferase (ALAT) and/or aspartate amino transferase (ASAT) >2 x upper normal serum levels)
* Anaemia
* Acute or chronic pancreatitis
* Struma or thyroid cancer
* Pregnancy or breast feeding
* Inability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
PASI (psoriasis area and severity index) | Baseline and after 2 months
DLQI (dermatology life quality index) | Baseline and after 2 months

SECONDARY OUTCOMES:
Body mass index | Baseline and after 2 months
CRP | Baseline and after 2 months
Skin biopsies | Baseline and after 2 months

CONTACTS AND LOCATIONS:
Overall Officials: AnneSofie Faurschou, MD PhD, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark